CLINICAL TRIAL: NCT02966015
Title: Product Evaluation of a Newly Developed Intermittent Catheter.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CP268
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Incontinence, Urinary
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Testing the new Coloplast Test catheter (Experimental): The subjects used the new Coloplast Test catheter for 1 week
  Interventions: Device: Coloplast test catheter

INTERVENTIONS:
Device: Coloplast test catheter — This is a newly developed catheter

SUMMARY:
The aim of the study is to investigate the navigation of a newly developed catheter.

ELIGIBILITY:
Inclusion Criteria:

1. Male and at least 18 years
2. Has used Intermittent self-catheterization at least 3 months
3. Has normal to slightly reduced hand mobility
4. Use catheter size CH12 or CH14 (must use same size during product evaluation)

Exclusion Criteria:

1. Currently receiving treatment for urinary tract infection
2. Currently receiving chemotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2016-05; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camilla F Vibjerg, Msc, Study Chair — Head of clinical operation

RESULTS

PARTICIPANT FLOW:
Groups:
- Tiemann/Coudé Users: The Tiemann/Coudé users used the new Coloplast Test catheter for 1 week. At inclusion the subjects were introduced to the product. They were asked to perform catheterization with Coloplast Test catheter. Those who were able to catheterize and wished to participate were included in the 1 week trial.
  Coloplast test catheter: This is a newly developed catheter
- Traditional Sleeve Catheter Users: The traditional sleeve catheter users used the new Coloplast Test catheter for 1 week. At inclusion the subjects were introduced to the product. They were asked to perform catheterization with Coloplast Test catheter. Those who were able to catheterize and wished to participate were included in the 1 week trial.
Period: Inclusion Visit
Arm/Group | Tiemann/Coudé Users | Traditional Sleeve Catheter Users
Started | 95 | 58
Completed | 87 | 55
Not Completed | 8 | 3
Not completed — did not answer questionnaire | 8 | 3
Period: Test Period
Arm/Group | Tiemann/Coudé Users | Traditional Sleeve Catheter Users
Started | 87 | 55
Completed | 87 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All the subjects enrolled in the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiemann/Coudé Users | Traditional Sleeve Catheter Users | Total
Number analyzed (Participants) | 95 | 58 | 153
Age, Customized [Number; unit: participants]
  Participants older than 18 years | 95 | 58 | 153
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 95 | 58 | 153

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Successfully Able to Insert Catheter
Description: The subjects had to evaluate if it was possible to insert and navigate the Coloplast Test catheter through urethra by the 5-point Likert question: "How did you find the catheter navigates through the urethra during insertion" ( Very easily, Easily, Neither/nor, Difficultly, Very difficultly, Not possible). The catheterization was considered successful if it was possible to insert the catheter, meaning that ifthey selected any other answer than 'not possible'.
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Tiemann/Coudé Users | Traditional Sleeve Catheter Users
Number analyzed (Participants) | 95 | 58
Participants | 82 | 58

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the trial period
Arm/Group | Tiemann/Coudé Users | Traditional Sleeve Catheter Users
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/58
Other Adverse Events (participants affected / at risk) | 0/95 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less